CLINICAL TRIAL: NCT01254669
Title: A Randomized Clinical Trial To Improve HPV Immunization in Haitian and African American Girls
Brief Title: An Intervention Study To Improve Human PapillomaVirus ( HPV) Immunization in Haitian and African American Girls
Acronym: HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Natalie Pierre-Joseph, Assistant Professor, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H26306
Record Dates: First submitted 2010-07-28; First posted 2010-12-06 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Cervical Cancer
Keywords: Haitian girls, African American girls; Brief Negotiated Interview; cognitive behavioral intervention; HPV vaccine; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control, standard of care (No Intervention): Mothers assigned to the Control Group received the low-literacy, standard-practice, HPV-vaccine information sheet
- BNI-brief Negotiated Interview (Experimental): The BNI intervention addressed mothers' beliefs, values, and concerns about HPV prevention and takes their priorities for health and well-being into account.
  Interventions: Behavioral: BNI-brief Negotiated Interview

INTERVENTIONS:
Behavioral: BNI-brief Negotiated Interview — use of a cognitive behavioral intervention to improve uptake of HPV vaccine
  Other Names: brief intervention to improve HPV vaccine in girls
  Arms: BNI-brief Negotiated Interview

SUMMARY:
In the United States, Black women are more likely to die of cervical cancer than White women. In developing countries and globally, Haitian immigrant women are more likely to die of cervical cancer than any other women in the world. Studies have shown a disparity in parental acceptance of the HPV vaccine with parents of Black adolescent girls being less likely to accept and comply with HPV immunization schedules than Whites. The objective of this study is to increase HPV immunization rates in Haitian and African American adolescent girls. The investigator's hypothesis is that a validated behavior change mechanism, brief-negotiating interviewing (BNI), will effectively increase the proportion of mothers who give consent for their daughters' HPV vaccine, which will ultimately lead to higher vaccination rates, and increase knowledge of HPV infection and the vaccine in Haitian immigrant and African American mothers.

DETAILED DESCRIPTION:
In the U.S., Black women have higher rates of cervical cancer than White women. Women in Haiti and Haitian immigrant women have among the highest rates of cervical cancer in the world. The recent introduction of the HPV vaccine provides an opportunity to reduce the disparity in cervical cancer rates between White and Black non-White (Haitians and US born African-Americans (AA)). Unfortunately, females ages 11-14 have low rates, 25%, of HPV vaccination. For the vaccine to be effective it must be given prior to the onset of sexual activity. Parents are a central audience for interventions to promote HPV vaccine uptake in children < 18 since parents have to consent.

Hypothesis: The objective of this study is to increase HPV immunization rates in Haitian and African American adolescent girls. My hypothesis is that a validated behavior change mechanism, brief-negotiating interviewing (BNI), will effectively increase the proportion of mothers who give consent for their daughters' HPV vaccine, which will ultimately lead to higher vaccination rates, and increase knowledge of HPV infection and the vaccine in Haitian immigrant and African American mothers.

Specific Aim 1a: Develop a script that will use BNI to address low-income Haitian immigrant and African American mothers' concern about HPV immunization

Specific Aim 1b: Teach community health workers to use BNI to enhance HPV acceptability Specific aim 2: Conduct a pilot, randomized clinical trial to determine feasibility effectiveness of BNI, and to obtain empirical estimates of study parameters to assess logistical aspects of a larger Randomized Clinical Trial (RCT). This will include assessing recruitment and retention of subjects, intervention delivery, and effect size.

Study design: The primary study design will be a RCT which will follow the CONSORT requirements for data reporting and analysis. One-hundred immigrant Haitian mothers bringing their adolescent daughters (age range 11 to 15) to clinic for routine care will be randomized to BNI (n=80) or to standard care (N=80) information about HPV vaccine). The primary outcome will be receipt of the first HPV vaccination in the adolescent within 1 month of randomization. The secondary outcome will be maternal knowledge about HPV vaccine. This study will provide key estimates so that we can conduct a fully-powered RCT, which will include completion of the primary HPV series (3 vaccinations) as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* 11-15 HPV vaccine eligible adolescent girls

Exclusion Criteria:

* Prior receipt of the HPV vaccine
* pregnant

Ages: 11 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: natalie joseph, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 100 English- and 100 Haitian Creole-speaking mothers of adolescent girls between April 2011 and September 2013 at the medical clinic ( pediatrics and adolescent clinic). Of 1,703 mothers approached during the study period,1,201 were ineligible. Of the 502 eligible, 302 declined and 200 (40%) were recruited &consented to pilot trial.
Pre-assignment Details: Following participant enrollment, but prior to group assignment, no significant event occurred. However, in our study after being randomized, participants provided demographic data. During data collection, one participants was excluded/self-withdrew from the trial for fear that demographic data may affect her immigration status/not documented.
Groups:
- Standard of Care: A clinical Pilot trials of a Brief Negotiated Intervention (a brief modified version of Motivational interview using a client-centered style) with mothers to improve Human Papilloma Virus (HPV) vaccination in Haitian and African-American adolescent daughters/girls compare to standard of care.
  Mothers assigned to the Control Group received the low-literacy, standard-practice, HPV vaccine information sheet usually given to all patients prior to vaccination. Control mothers met once with the research assistant to collect demographic characteristics, HPV knowledge, and vaccine status of the daughter on the day of visit. No Brief Negotiated Intervention (BNI) counseling was provided.
- Brief Negotiated Inteview (BNI) Intervention: A clinical Pilot trials of a Brief Negotiated Intervention (a brief modified version of Motivational interview using a client-centered style) with mothers to improve HPV vaccination in Haitian and African-American adolescent daughters/girls compare to standard of care.
  One hundred mothers received intervention (n=50 Haitian, 50 African-American). Four Haitian mothers did not receive intervention because (i) One was called to see the clinical provider during the intervention and did not return (n=1), and (ii) time constraints (n=2) and one dropped out for fear information from study will affect her immigration status
Period: Overall Study
Arm/Group | Standard of Care | Brief Negotiated Inteview (BNI) Intervention
Started | 100 | 100
Completed | 97 | 96
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — time constraint | 2 | 2
Not completed — called to clinic during intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: A clinical Pilot trials of a Brief Negotiated Intervention (a brief modified version of Motivational interview using a client-centered style) with mothers to improve HPV vaccination in Haitian and African-American adolescent daughters/girls compare to standard of care.
  Of the 100 women in the Control Group (n=50 Haitian, 50 African-American), three African-American mothers did not complete Control Group activities because they did not complete the survey. Reasons for initial dropout/decline to participate included being too busy, not interested, time constraints, and daughter not sexually active upon hearing study has to do with HPV vaccine.
- BNI/Intervention: One hundred mothers received intervention (n=50 Haitian, 50 African-American). Four Haitian mothers did not receive intervention because (i) One was called to see the clinical provider during the intervention and did not return (n=1), and (ii) time constraints (n=2), one for immigration status .
- Total: Total of all reporting groups
Arm/Group | Standard of Care | BNI/Intervention | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 41 (7) | 40 (9) | 41 (8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 100 | 100 | 200
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 100 | 100 | 200
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
knowledge of HPV vaccine [Mean (Standard Deviation); unit: units on a scale] — Assessment of HPV knowledge range from 0 (minimal) to 12 ( maximal knowledge)
  units on a scale | 5 (4) | 6 (4) | 5 (4)

OUTCOME MEASURES:

1. Primary Outcome: The Receipt of the First HPV Vaccination
Description: Receipt of the first HPV vaccination among adolescent daughters of the participants
Time Frame: within 1 month of randomization
Population: The number of participants for analysis was determined based on number of participants enrolled and who answered questions of interest.
Measure: Number; unit: percentage of participants
Groups:
- Standard of Care: A clinical Pilot trials of a Brief Negotiated Intervention (a brief modified version of Motivational interview using a client-centered style) with mothers to improve HPV vaccination in Haitian and African-American adolescent daughters/girls compare to standard of care.
  Of the 100 women in the Control Group (n=50 Haitian, 50 African-American), received the standard of care handout given to patients on the vaccine they will be getting that day. three African-American mothers did not complete Control Group activities because they did not complete the survey. Reasons for initial dropout/decline to participate included being too busy, not interested, time constraints, and daughter not sexually active upon hearing study has to do with HPV vaccine.
- BNI/Intervention: Intervention was administered to 100 African-American and Haitian mothers over 10-20 minutes prior to seeing the health provider if the daughter had never received the HPV vaccine, or after seeing the health provider if the daughter did not received the vaccine during the visit.
Arm/Group | Standard of Care | BNI/Intervention
Number analyzed (Participants) | 97 | 96
percentage of participants | 51 | 56

2. Secondary Outcome: The Secondary Outcome Will be Maternal Knowledge About HPV Vaccine.
Description: post-educational intervention assessment of HPV knowledge ranges from 0 (minimal knowledge) to 12 (maximal knowledge)
Time Frame: 1 hour after intervention
Population: The number of participants for analysis was determined based on the total enrolled and who responded to knowledge questions
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- BNI Post-educational Intervention Group: A clinical Pilot trials of a Brief Negotiated Intervention (a brief modified version of Motivational interview using a client-centered style) with mothers to improve HPV vaccination in Haitian and African-American adolescent daughters/girls compare to standard of care.
  Post-educational interventional assessment of HPV knowledge ranges from 0(minimal knowledge) to 12 (maximal knowledge)
- Control Group: Did not receive any BNI intervention on the pre and post measure
Arm/Group | BNI Post-educational Intervention Group | Control Group
Number analyzed (Participants) | 99 | 96
units on a scale | 10 (2) | 5 (2)

ADVERSE EVENTS:
Time Frame: 1 year- no adverse event over
Description: no adverse event
Groups:
- BNI/Intervention: One hundred mothers received intervention (n=50 Haitian, 50 African-American). . Four Haitian mothers did not receive intervention because (i) One was called to see the clinical provider during the intervention and did not return (n=1), and (ii) time constraints (n=2), one due to fear of information affecting immigration status.
Arm/Group | Standard of Care | BNI/Intervention
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

LIMITATIONS AND CAVEATS:
Limitations:small sample,Enrolling only mothers, of daughters who are African-American and Haitians lead to longer recruitment time/non-generalizable data. Future studies should include heterogeneous ethnicities,fathers, sons, and any legal guardian.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No